CLINICAL TRIAL: NCT00496834
Title: A Randomized, Open-label, Comparative, Non-inferiority, Multicenter Study to Compare Efficacy of Losartan Potassium Group and Carvedilol Group on Arterial Stiffness in Essential Hypertension Patients
Brief Title: LAAS (Losartan Anti-Atherosclerosis Study)(0954-330)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954-330; 2007_015; NCT01001416 (obsolete NCT alias)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Hydrochlorothiazide

ARMS (2):
- 1 (Experimental): Losartan or Losartan/HCTZ
  Interventions: Drug: losartan potassium; Drug: Comparator: losartan (+) hydrochlorothiazide (HCTZ)
- 2 (Active Comparator): Carvedilol or Carvedilol/HCTZ
  Interventions: Drug: Comparator: carvedilol; Drug: Comparator: carvedilol (+) hydrochlorothiazide

INTERVENTIONS:
Drug: losartan potassium — Once daily , Cozaar® (losartan) 50 mg, Cozaar® (losartan) 100 mg, Cozaar Plus®-pro Tab. (losartan 100 mg/ hydrochlorothiazide 12.5 mg) or Cozaar Plus®-F Tab. (losartan 100 mg / hydrochlorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan)
  Arms: 1
Drug: Comparator: carvedilol — Once daily, Dilatrend Tab® (carvedilol) 12.5 mg, Dilatrend Tab® (carvedilol) 25 mg, Dilatrend Tab® (carvedilol) 25 mg plus half Dichlozid Tab® (hydrochlorothiazide 25 mg) or Dilatrend Tab® (carvedilol) 25 mg plus full Dichlozid Tab® (hydrochlorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan)
  Arms: 2
Drug: Comparator: losartan (+) hydrochlorothiazide (HCTZ) — Once daily , Cozaar® (losartan) 50 mg, Cozaar® (losartan) 100 mg, Cozaar Plus®-pro Tab. (losartan 100 mg/ hydrochlorothiazide 12.5 mg) or Cozaar Plus®-F Tab. (losartan 100 mg / hydrochlorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan)
  Arms: 1
Drug: Comparator: carvedilol (+) hydrochlorothiazide — Once daily, Dilatrend Tab® (carvedilol) 12.5 mg, Dilatrend Tab® (carvedilol) 25 mg, Dilatrend Tab® (carvedilol) 25 mg plus half Dichlozid Tab® (hydrochlorothiazide 25 mg) or Dilatrend Tab® (carvedilol) 25 mg plus full Dichlozid Tab® (hydrochlorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan)
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate efficacy, arterial stiffness measured by Pulse Wave Velocity (PWV) of Losartan potassium group compared to Carvedilol group after 24 weeks of treatment in patients with the essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female adults, 18 years or over
* Essential Hypertension with mean SBP (systolic blood pressure) ≥ 140 mm Hg or mean DBP (diastolic blood pressure) ≥ 90 mm Hg* when blood pressure is measured at Visit 1(week -2) and at Visit 2(week 0).

If diabetes patients, mean SBP ≥ 130 mm Hg or mean DBP ≥ 80 mm Hg (Mean of blood pressure values measured consecutively at least 2 minutes apart)

* Patient who is willing to, and is able to sign the informed consent form

Exclusion Criteria:

* Patient Is Pregnant Or Breastfeeding, Or Expecting To Conceive Within The Projected Duration Of The Study
* Patient Has Known Or Suspected Secondary Hypertension Of Any Etiology
* Patient has history of malignant hypertension
* Patient has history of cerebrovascular accident (cerebral infarction) or myocardiac infarction within the last 6 months
* Patient takes antihypertensive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2009-09-01 (Actual); Study Completion 2009-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 centers participated in this study (7 medical centers of university).
  FPE (First patient enrolled): Feb-2008, FPI (First patient in): Feb-2008, LPO (Last patient out): Sep-2009
Groups:
- Losartan: Once daily , Cozaar® (losartan) 50 mg, Cozaar® (losartan) 100 mg, Cozaar Plus®-pro Tab. (losartan 100 mg / hydrochrolorothiazide 12.5 mg) or Cozaar Plus®-F Tab. (losartan 100 mg / hydrochrolorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan).
- Carvedilol: Once daily, Dilatrend Tab® (carvedilol) 12.5 mg, Dilatrend Tab® (carvedilol) 25 mg, Dilatrend Tab® (carvedilol) 25 mg plus half Dichlozid Tab® (hydrochlorothiazide 25 mg) or
  Dilatrend Tab® (carvedilol) 25 mg plus full Dichlozid Tab® (hydrochlorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan).
Period: Overall Study
Arm/Group | Losartan | Carvedilol
Started | 101 | 100
Completed | 83 | 87
Not Completed | 18 | 13
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Contraindicated medication administered | 0 | 1
Not completed — Inclusion/exclusion criteria not met | 3 | 2
Not completed — Adverse Event | 5 | 3
Not completed — IP administration violation | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Blood Pressure control failure | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Carvedilol | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (9.3) | 50.1 (10.2) | 49.6 (9.7)
Age, Customized [Number; unit: participants]
  >= 18 to < 65 years | 96 | 91 | 187
  >=65 years | 5 | 9 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 57 | 120
  Male | 38 | 43 | 81
DBP (diastolic blood pressure) [Mean (Standard Deviation); unit: mm Hg] | 96.4 (8.8) | 96.4 (8.3) | 96.4 (8.5)
Height [Mean (Standard Deviation); unit: Centimeters] | 164.9 (7.8) | 163.3 (9.2) | 164.1 (8.5)
PWV (pulse wave velocity) [Mean (Standard Deviation); unit: meters/second] | 7.6 (1.4) | 7.7 (1.4) | 7.6 (1.4)
Pulse [Mean (Standard Deviation); unit: BPM (beats per minute)] | 71.8 (10.0) | 72.3 (10.0) | 72.0 (10.0)
SBP (systolic blood pressure) [Mean (Standard Deviation); unit: mm Hg] | 150.6 (11.0) | 152.7 (12.1) | 151.6 (11.6)
Weight [Mean (Standard Deviation); unit: Kilograms] | 70.9 (10.6) | 69.9 (13.2) | 70.4 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Pulse Wave Velocity (PWV) Changes From Baseline (Visit 2) to 24 Weeks (Visit 6) After the Administration of the Study Drug
Description: Analysis was performed in the modified intention to treat (mITT) population.
Time Frame: Baseline and 24 Weeks
Population: Participants for analysis was modified intention to treat (Number of patients: Losartan group was 88, Carvedilol group was 94). Missing data were imputed by the last observation carried forward (LOCF) technique.
Measure: Mean (Standard Deviation); unit: meters/second
Groups:
- Losartan: Once daily , Cozaar® (losartan) 50 mg, Cozaar® (losartan) 100 mg, Cozaar Plus®-pro Tab. (losartan 100 mg / hydrochrolorothiazide 12.5 mg) or Cozaar Plus®-F Tab. (losartan 100 mg / hydrochrolorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan) and patients who 1) had baseline measurements before randomization, 2) had taken the study drug more than once after randomization, 3) had one measurement after the initiation of the administration and 4) did not commit major violation.
- Carvedilol: Once daily, Dilatrend Tab® (carvedilol) 12.5 mg, Dilatrend Tab® (carvedilol) 25 mg, Dilatrend Tab® (carvedilol) 25 mg plus half Dichlozid Tab® (hydrochlorothiazide 25 mg) or
  Dilatrend Tab® (carvedilol) 25 mg plus full Dichlozid Tab® (hydrochlorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan) and patients who 1) had baseline measurements before randomization, 2) had taken the study drug more than once after randomization, 3) had one measurement after the initiation of the administration and 4) did not commit major violation.
Arm/Group | Losartan | Carvedilol
Number analyzed (Participants) | 88 | 94
meters/second | 0.28 (1.29) | -0.12 (1.55)
Statistical Analysis 1: Comparison: Losartan vs Carvedilol; Participants for analysis was modified intention to treat (Number of patients: Losartan group was 88, Carvedilol group was 94); Test type: Non-Inferiority or Equivalence — non-inferiority margin= -1.5m/s; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.83 to 0.01], Standard Deviation 1.43 — The lower limit of ≥-1.5m/s was judged to prove the non-inferiority of the test group to the control group

2. Primary Outcome: PWV Changes From Baseline (Visit 2) to 24 Weeks (Visit 6) After the Administration of the Study Drug
Description: Analysis was performed in the per protocol (PP) population which additionally excludes certain protocol violations as described in the analysis plan.
Time Frame: Baseline and 24 Weeks
Population: Participants for analysis was per protocol (Number of patients: Losartan group was 54, Carvedilol group was 67). Missing data were imputed by the last observation carried forward (LOCF) technique. For the primary efficacy endpoints, Per protocol analysis approach was supplementary used.
Measure: Mean (Standard Deviation); unit: meters/second
Groups:
- Losartan: Once daily , Cozaar® (losartan) 50 mg, Cozaar® (losartan) 100 mg, Cozaar Plus®-pro Tab. (losartan 100 mg / hydrochrolorothiazide 12.5 mg) or Cozaar Plus®-F Tab. (losartan 100 mg / hydrochrolorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan) and patients who 1) had baseline measurements before randomization, 2) had taken the study drug more than once after randomization, 3) had one measurement after the initiation of the administration 4) did not commit major violation and 5) did not have protocol violation including erroneous prescription of the investigational drug, baseline PWV test date violation, PWV test date violation 24 weeks after the administration of the investigational drug, titration violation, use of prohibited concomitant drugs, visit window violation and inclusion/exclusion criteria violation.
- Carvedilol: Once daily, Dilatrend Tab® (carvedilol) 12.5 mg, Dilatrend Tab® (carvedilol) 25 mg, Dilatrend Tab® (carvedilol) 25 mg plus half Dichlozid Tab® (hydrochlorothiazide 25 mg) or
  Dilatrend Tab® (carvedilol) 25 mg plus full Dichlozid Tab® (hydrochlorothiazide 25 mg), 24 weeks (Patients who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan) and patients who 1) had baseline measurements before randomization, 2) had taken the study drug more than once after randomization, 3) had one measurement after the initiation of the administration 4) did not commit major violation and 5) did not have protocol violation including erroneous prescription of the investigational drug, baseline PWV test date violation, PWV test date violation 24 weeks after the administration of the investigational drug, titration violation, use of prohibited concomitant drugs, visit window violation and inclusion/exclusion criteria violation.
Arm/Group | Losartan | Carvedilol
Number analyzed (Participants) | 54 | 67
meters/second | 0.16 (1.25) | -0.20 (1.50)
Statistical Analysis 1: Comparison: Losartan vs Carvedilol; Participants for analysis was per protocol (Number of patients: Losartan group was 54, Carvedilol group was 67). For the primary efficacy endpoints, Per protocol analysis approach was supplementary used; Test type: Non-Inferiority or Equivalence — non-inferiority margin=-1.5m/s; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.86 to 0.15], Standard Deviation 1.40 — The lower limit of ≥-1.5m/s was judged to prove the non-inferiority of the test group to the control group

3. Secondary Outcome: Systolic Blood Pressure (SBP) Mean Changes From Baseline (Visit 2) to 24 Weeks (Visit 6) After the Administration of the Study Drug
Time Frame: Baseline and 24 weeks
Population: Participants for analysis was modified intention to treat (Number of patients: Losartan group was 88, Carvedilol group was 94) Missing data were imputed by the last observation carried forward (LOCF) technique.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan | Carvedilol
Number analyzed (Participants) | 88 | 94
mm Hg | -15.08 (14.59) | -14.81 (15.38)
Statistical Analysis 1: Comparison: Losartan vs Carvedilol; Test type: Superiority or Other; p = 0.9032, t-test, 2 sided — Significance level=0.05; The secondary efficacy analysis was performed in the modified intention to treat population using t-test

4. Secondary Outcome: Diastolic Blood Pressure (DBP) Mean Changes From Baseline (Visit 2) to 24 Weeks (Visit 6) After the Administration of the Study Drug
Time Frame: Baseline and 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan | Carvedilol
Number analyzed (Participants) | 88 | 94
mm Hg | -8.43 (9.29) | -7.81 (9.61)
Statistical Analysis 1: Comparison: Losartan vs Carvedilol; Test type: Superiority or Other; p = 0.6574, t-test, 2 sided — Significance level=0.05; The secondary efficacy analysis was performed in the modified intention to treat population using t-test

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from first administration of study drug up to 14 days after the administration of final dose.
Groups:
- Losartan: Once daily , Cozaar® (losartan) 50 mg, Cozaar® (losartan) 100 mg, Cozaar Plus®-pro Tab. (losartan 100 mg / hydrochrolorothiazide 12.5 mg) or Cozaar Plus®-F Tab. (losartan 100 mg / hydrochrolorothiazide 25 mg), 24 weeks (Subjects who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan) and patients who received the investigational drug at least more than once.
- Carvedilol: Once daily, Dilatrend Tab® (carvedilol) 12.5 mg, Dilatrend Tab® (carvedilol) 25 mg, Dilatrend Tab® (carvedilol) 25 mg plus half Dichlozid Tab® (hydrochlorothiazide 25 mg) or
  Dilatrend Tab® (carvedilol) 25 mg plus full Dichlozid Tab® (hydrochlorothiazide 25 mg), 24 weeks (Subjects who have failed in blood pressure control, increase the study medication dose step by step according to the titration plan) and patients who received the investigational drug at least more than once.
Arm/Group | Losartan | Carvedilol
Serious Adverse Events (participants affected / at risk) | 5/101 | 6/100
Other Adverse Events (participants affected / at risk) | 35/101 | 51/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=101) | Carvedilol (N=100)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=101) | Carvedilol (N=100)
Headache (Nervous system disorders) | 8 (8) | 9 (12)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 7 (10)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 3 (3)
Chest discomfort (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Face oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.